CLINICAL TRIAL: NCT03295318
Title: A Phase 2, Observer-blind, Randomized, Controlled Study to Evaluate the Safety and Immunogenicity of Two Formulations of Investigational Meningococcal Groups ACYWX Conjugate Vaccine, Administered to Healthy Malian Children 12-16 Months of Age
Brief Title: Clinical Study of Meningococcal ACYWX Conjugate Vaccine, in 12-16 Month Olds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACYWX-002; CVIA-058 (Other: PATH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-27 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2021-08

CONDITIONS: Meningitis, Meningococcal
Keywords: Neisseria meningitidis; conjugate meningococcal vaccine; meningococcal serogroup X
MeSH Terms: conditions — Meningitis, Meningococcal | interventions — Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind wherein the pharmacist and other study staff involved in vaccine administration will be aware of the treatment allocation.
  The other study staff involved in safety assessments will be masked to treatment arm. The laboratory involved in immunogenicity analysis will also be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adjuvanted study formulation NmCV-5 (Experimental): Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Interventions: Biological: Adjuvanted study formulation NmCV-5
- Non-adjuvanted study formulation NmCV-5 (Experimental): Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Interventions: Biological: Non-adjuvanted study formulation NmCV-5
- Menactra (Active Comparator): Subjects in this arm will licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Interventions: Biological: Menactra

INTERVENTIONS:
Biological: Non-adjuvanted study formulation NmCV-5 — Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
  Other Names: MenACYWX
  Arms: Non-adjuvanted study formulation NmCV-5
Biological: Adjuvanted study formulation NmCV-5 — Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
  Other Names: Adj MenACYWX
  Arms: Adjuvanted study formulation NmCV-5
Biological: Menactra — Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
  Other Names: MenACYW-D
  Arms: Menactra

SUMMARY:
Out of the 13 identified serogroups of Neisseria meningitidis (Nm) the six serogroups (A, B, C, W, Y and X) are responsible for majority of infections. Presently available vaccines effectively protect against A, B, C, W and Y serogroups; but no vaccine that is protective against serogroup X is available yet.

Serum Institute of India Private Limited (SIIPL) has developed a conjugate vaccine against serogroups A, C, Y, W and X (NmCV-5).

The first-in-human Phase 1 study was among 60 healthy adults in USA did not show no any safety issues.

This phase 2 study is designed to evaluate safety and immunogenicity of the non-adjuvanted and adjuvanted formulations of NmCV-5 in healthy children 12-16 months of age, in comparison with the licensed quadrivalent meningococcal conjugate vaccine (Menactra®).

Both vaccines will be administered in two dose schedule 3 months apart. among vaccine-naïve healthy subjects in Mali. Safety will be assessed by collecting solicited reactions till day 7 post each dose whereas adverse events will be collected throughout the study. Each subject will be followed up for 84 days post each vaccine dose.

The vaccine immunogenicity will measured using a rabbit complement serum bactericidal activity assay (rSBA).

ELIGIBILITY:
Inclusion Criteria:

* Male and female children between 12 months and 16 months old inclusive (minimum 365 days of age and maximum 16 months plus 29 days of age);
* For whom parent(s)/legal guardian(s) have given written informed consent after the nature of the study has been explained according to local regulatory requirements;
* Who the investigator believes that their parent(s)/ guardian(s) will be available for all the subject visits and would comply with the requirements of the protocol (e.g., timely reporting of adverse events, availability for study site visits and home visits);
* Individuals in good health as determined by the outcome of medical history, physical examination and clinical judgment of the investigator.
* Individuals who completed their local infant EPI schedule through 9 months of age (except MenAfriVac dose). A birth dose of OPV is not required)

Exclusion Criteria:

* History of any meningococcal vaccine administration.
* Current or previous, confirmed or suspected disease caused by N. meningitidis.
* Household contact with and/or intimate exposure to an individual with any laboratory confirmed N. meningitidis infection within 60 days of enrolment.
* History of severe allergic reactions after previous vaccinations or hypersensitivity to any study vaccine component including tetanus, diphtheria and diphtheria toxoid (CRM197).
* Acute or chronic, clinically significant pulmonary, cardiovascular, metabolic, neurological, hepatic, or renal functional abnormality, as determined by medical history or physical examination.
* Any confirmed or suspected condition with impaired/altered function of immune system (immunodeficient or autoimmune conditions).
* Have any bleeding disorder which is considered as a contraindication to intramuscular injection or blood draw.
* Severe acute malnutrition.
* A family history of congenital or hereditary immunodeficiency.
* History of either hepatitis B or hepatitis C virus infection or human immunodeficiency virus infection.
* Major congenital defects.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within three months prior to the study vaccination or planned use throughout the study period. (For corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg per day. Inhaled, intranasal and topical steroids are allowed).
* Administration of blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation in the past 3 months or planned use throughout the study period.
* Administration of any vaccine within 28 days prior to enrolment in the study or planned administration of any vaccine within 14 days before or after any study vaccination.
* Use of any investigational or non-registered drug or vaccine within 30 days prior to the administration of study vaccines or planned during the study.
* Malaria infection as confirmed by a Rapid Diagnostic Test.
* Individuals who are close family members of individuals conducting this study.
* Have experienced a moderate or severe acute infection and/or fever (defined as temperature ≥ 37.5°C) within 3 days prior to enrolment.
* Have received systemic antibiotic treatment within 3 days prior to enrolment.
* Non-residence in the study area or intent to move out within six months.
* Any condition which, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study

Ages: 12 Months to 16 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 375 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre pour le Développement des Vaccins du Mali, ex-Institut Marchoux, Ministry of Health, BP251, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tapia MD, Sow SO, Naficy A, Diallo F, Haidara FC, Chaudhari A, Martellet L, Traore A, Townsend-Payne K, Borrow R, Hosken N, Smolenov I, Pisal SS, LaForce FM, Dhere RM, Kapse D, Tang Y, Alderson MR, Kulkarni PS. Meningococcal Serogroup ACWYX Conjugate Vaccine in Malian Toddlers. N Engl J Med. 2021 Jun 3;384(22):2115-2123. doi: 10.1056/NEJMoa2013615. PMID 34077644

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 515 toddlers were consented to withhold Mali EPI MenAfriVac vaccination at 9 months and were invited to return at 12 months for a second consent and final eligibility assessment. Among these, 136 were subsequently not consented, of which 127 received MenAfriVac to align with their EPI schedule. 379 participants were subsequently consented and assessed for eligibility, of which 2 did not meet eligibility criteria and 1 withdrew consent prior to randomization, leading to 376 randomized.
Groups:
- Non-adjuvanted Study Formulation NmCV-5: Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Non-adjuvanted study formulation NmCV-5: Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
- Adjuvanted Study Formulation NmCV-5: Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Adjuvanted study formulation NmCV-5: Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
- Menactra: Subjects in this arm will licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Menactra: Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
Period: Overall Study
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Started | 150 | 150 | 76
Received First Vaccination | 149 (1 subject withdrew consent after randomization, but prior to vaccination.) | 150 | 76
Received Second Vaccination | 144 | 145 | 73
Completed | 144 | 145 | 71
Not Completed | 6 | 5 | 5
Not completed — Withdrawal by Subject prior to initial vaccination | 1 | 0 | 0
Not completed — Death | 1 | 1 | 1
Not completed — Protocol Violation | 4 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Subject discontinued due to travel | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra | Total
Number analyzed (Participants) | 149 | 150 | 76 | 375
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.1 (0.60) | 12.1 (0.53) | 12.1 (0.44) | 12.1 (0.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 68 | 36 | 177
  Male | 76 | 82 | 40 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 149 | 150 | 76 | 375
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 149 | 150 | 76 | 375
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Length (cm) [Mean (Standard Deviation); unit: centimeters] | 72.94 (2.533) | 73.03 (2.858) | 72.59 (2.460) | 72.91 (2.652)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 8.81 (1.002) | 8.89 (1.140) | 8.77 (1.007) | 8.83 (1.059)
Temperature (°C) [Mean (Standard Deviation); unit: Celsius] | 36.25 (0.266) | 36.24 (0.299) | 36.24 (0.270) | 36.25 (0.279)
Heart Rate (beats/min) [Mean (Standard Deviation); unit: Beats/minute] | 110.8 (5.80) | 111.3 (5.74) | 110.8 (6.09) | 111.0 (5.83)
Respiratory Rate (breaths per minute) [Mean (Standard Deviation); unit: Breaths per minute] | 31.8 (3.00) | 31.7 (2.67) | 32.6 (3.05) | 31.9 (2.89)

OUTCOME MEASURES:

1. Primary Outcome: Severe Solicited Adverse Event
Description: Number and Percentage of subjects with at least one severe solicited AE within 7 days after any study vaccination (Days 0-6 and Days 84-90)
Time Frame: 7 days post each vaccination
Population: Analysis population different for severe solicited AEs within 7 days after 2nd study vaccination, as number of subjects who received the 2nd dose was less than those that received the first dose. Reasons outlined in Participant Flow.
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Adjuvanted Study Formulation NmCV-5 | Non-adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 149 | 150 | 76
participants
  Number of subjects with at least one severe solicited AE reported within 7 days after 1st dose | 0 [0.00 to 2.45] | 0 [0.00 to 2.43] | 0 [0.00 to 4.74]
  Number of subjects with at least one severe solicited AE reported within 7 days after 2nd dose: number analyzed (Participants) | 144 | 145 | 73
  Number of subjects with at least one severe solicited AE reported within 7 days after 2nd dose | 0 [0.00 to 2.53] | 0 [0.00 to 2.51] | 0 [0.00 to 4.93]

2. Secondary Outcome: Seroprotective rSBA Titres
Description: Percentage of subjects with rSBA titer ≥ 8 against serogroups A, C, W, Y and X at Visits Day 0 (Baseline), Day 28 (28 days after dose 1), Day 84 (prior to dose 2) and Day 112 (28 days after dose 2)
Time Frame: 112 days
Population: per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 144 | 144 | 72
Participants
  Serogroup A Day 0 | 16 | 19 | 10
  Serogroup A Day 28 | 144 | 144 | 71
  Serogroup A Day 84 | 144 | 144 | 71
  Serogroup A Day 112 | 144 | 144 | 72
  Serogroup C Day 0 | 3 | 0 | 0
  Serogroup C Day 28 | 143 | 143 | 56
  Serogroup C Day 84 | 141 | 139 | 51
  Serogroup C Day 112 | 144 | 144 | 72
  Serogroup W Day 0 | 9 | 6 | 2
  Serogroup W Day 28 | 142 | 141 | 65
  Serogroup W Day 84 | 140 | 142 | 59
  Serogroup W Day 112 | 144 | 144 | 72
  Serogroup X Day 0 | 15 | 12 | 6
  Serogroup X Day 28 | 144 | 143 | 15
  Serogroup X Day 84 | 144 | 143 | 14
  Serogroup X Day 112 | 143 | 144 | 25
  Serogroup Y Day 0 | 17 | 21 | 10
  Serogroup Y Day 28 | 141 | 143 | 64
  Serogroup Y Day 84 | 141 | 143 | 65
  Serogroup Y Day 112 | 144 | 144 | 71

3. Secondary Outcome: Long Term Protective rSBA Titres
Description: Percentage of subjects with rSBA titer ≥ 128 against serogroups A, C, W, Y and X at Visits Day 0, Day 28, Day 84 and Day 112
Time Frame: 112 days
Population: Per Protocol Population
Measure: Count of Participants; unit: Participants
Groups:
- Menactra: Subjects in this arm will receive licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Menactra: Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 144 | 144 | 72
Participants
  Serogroup A Day 0 | 16 | 18 | 10
  Serogroup A Day 28 | 144 | 144 | 71
  Serogroup A Day 84 | 144 | 143 | 71
  Serogroup A Day 112 | 144 | 144 | 72
  Serogroup C Day 0 | 2 | 0 | 0
  Serogroup C Day 28 | 142 | 140 | 39
  Serogroup C Day 84 | 133 | 131 | 26
  Serogroup C Day 112 | 144 | 144 | 68
  Serogroup W Day 0 | 8 | 5 | 2
  Serogroup W Day 28 | 142 | 141 | 65
  Serogroup W Day 84 | 137 | 139 | 57
  Serogroup W Day 112 | 144 | 144 | 69
  Serogroup X Day 0 | 15 | 12 | 6
  Serogroup X Day 28 | 144 | 143 | 15
  Serogroup X Day 84 | 144 | 143 | 14
  Serogroup X Day 112 | 143 | 144 | 22
  Serogroup Y Day 0 | 16 | 21 | 10
  Serogroup Y Day 28 | 140 | 143 | 64
  Serogroup Y Day 84 | 138 | 141 | 60
  Serogroup Y Day 112 | 144 | 144 | 66

4. Secondary Outcome: Rise in rSBA Titres
Description: Percentage of subjects with fourfold rise in rSBA titers against serogroups A, C, W, Y and X at Visits Day 28 and Day 112.
  * For subjects with a pre-vaccination rSBA titer < 8, a post-vaccination titer of ≥ 32;
  * For subjects with a pre-vaccination rSBA titer ≥ 8, an increase in rSBA titer of at least 4 times the pre-vaccination titer
Time Frame: 112 days
Population: Per protocol population
Measure: Count of Participants; unit: Participants
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 144 | 144 | 72
Participants
  Serogroup A: Day 28 | 143 | 144 | 70
  Serogroup A: Day 112 | 143 | 144 | 71
  Serogroup C: Day 28 | 141 | 141 | 50
  Serogroup C: Day 112 | 142 | 144 | 72
  Serogroup W: Day 28 | 140 | 140 | 65
  Serogroup W: Day 112 | 142 | 143 | 71
  Serogroup X: Day 28 | 144 | 142 | 12
  Serogroup X: Day 112 | 143 | 143 | 19
  Serogroup Y: Day 28 | 140 | 142 | 63
  Serogroup Y: Day 112 | 144 | 142 | 71

5. Secondary Outcome: Geometric Mean of rSBA Titres
Description: rSBA GMT for serogroups A, C, W, Y and X at Visits Day 0, Day 28, Day 84 and Day 112
Time Frame: 112 Days
Population: Per protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean rSBA Titer
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 144 | 144 | 72
Geometric Mean rSBA Titer
  Serogroup A Day 0 | 3.8 [2.81 to 5.18] | 4.3 [3.08 to 5.89] | 4.4 [2.74 to 6.95]
  Serogroup A Day 28 | 7732.2 [6462.42 to 9251.52] | 7368.8 [6210.80 to 8742.81] | 3866.1 [2841.91 to 5259.43]
  Serogroup A Day 84 | 4687.0 [3919.72 to 5604.44] | 4488.3 [3600.74 to 5594.57] | 2786.9 [2003.18 to 3877.24]
  Serogroup A Day 112 | 6226.3 [5435.42 to 7132.33] | 6166.7 [5375.47 to 7047.35] | 4871.0 [3833.59 to 6189.12]
  Serogroup C Day 0 | 2.2 [1.97 to 2.37] | 2.0 [NA to NA] — *For Serogroup C, all subjects have same titer values at baseline in Adjuvanted NmCV-5 and MenACWY-D arms. | 2.0 [NA to NA] — *For Serogroup C, all subjects have same titer values at baseline in Adjuvanted NmCV-5 and MenACWY-D arms.
  Serogroup C Day 28 | 1143.9 [929.32 to 1407.98] | 1095.4 [877.66 to 1367.12] | 67.8 [39.69 to 115.84]
  Serogroup C Day 84 | 436.8 [342.33 to 557.34] | 348.4 [272.51 to 445.33] | 29.6 [18.73 to 46.87]
  Serogroup C Day 112 | 1366.9 [1173.58 to 1592.01] | 1393.4 [1200.54 to 1617.35] | 410.3 [324.93 to 518.11]
  Serogroup W Day 0 | 2.8 [2.22 to 3.52] | 2.5 [2.09 to 2.91] | 2.2 [1.91 to 2.64]
  Serogroup W Day 28 | 6533.4 [4868.00 to 8768.46] | 5363.2 [3927.83 to 7323.21] | 1127.5 [614.73 to 2067.93]
  Serogroup W Day 84 | 2555.6 [1839.63 to 3550.22] | 2222.6 [1673.59 to 2951.80] | 483.3 [242.96 to 961.24]
  Serogroup W Day 112 | 8035.8 [6255.62 to 10322.51] | 7056.4 [5622.17 to 8856.57] | 2482.8 [1567.27 to 3933.27]
  Serogroup X Day 0 | 3.5 [2.70 to 4.61] | 3.2 [2.50 to 4.19] | 3.2 [2.21 to 4.66]
  Serogroup X Day 28 | 7548.3 [6442.99 to 8843.32] | 8152.7 [6717.91 to 9893.84] | 6.9 [3.82 to 12.56]
  Serogroup X Day 84 | 3511.3 [2934.73 to 4201.08] | 3113.2 [2552.53 to 3796.93] | 6.7 [3.73 to 11.91]
  Serogroup X Day 112 | 5363.2 [4523.30 to 6359.15] | 6286.6 [5515.16 to 7165.86] | 11.6 [6.35 to 21.34]
  Serogroup Y Day 0 | 3.6 [2.74 to 4.64] | 4.1 [3.08 to 5.55] | 3.9 [2.63 to 5.86]
  Serogroup Y Day 28 | 2366.2 [1837.37 to 3047.14] | 3010.0 [2490.61 to 3637.74] | 676.9 [392.43 to 1167.54]
  Serogroup Y Day 84 | 1171.7 [891.95 to 1539.31] | 1386.8 [1129.10 to 1703.21] | 426.4 [252.21 to 720.93]
  Serogroup Y Day 112 | 3189.0 [2700.52 to 3765.84] | 3266.7 [2800.84 to 3810.01] | 1194.5 [809.00 to 1763.78]

6. Secondary Outcome: Solicited Reactions
Description: Solicited local and systemic AEs reported during the 7 days after each vaccination (Days 0-6 and Days 84-90);
Time Frame: 7 days post each vaccination
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Non-adjuvanted NmCV-5 (Days 0-6); Non-adjuvanted NmCV-5 (Days 84-90): Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by at least 84 days.
  Non-adjuvanted study formulation NmCV-5: Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysaccharide antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
- Adjuvanted NmCV-5 (Days 0-6); Adjuvanted NmCV-5 (Days 84-90): Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by at least 84 days.
  Adjuvanted study formulation NmCV-5: Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysaccharide antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
- Menactra (Days 0-6); Menactra (Days 84-90): Subjects in this arm will receive licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Menactra: Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
Arm/Group | Non-adjuvanted NmCV-5 (Days 0-6) | Adjuvanted NmCV-5 (Days 0-6) | Menactra (Days 0-6) | Non-adjuvanted NmCV-5 (Days 84-90) | Adjuvanted NmCV-5 (Days 84-90) | Menactra (Days 84-90)
Number analyzed (Participants) | 149 | 150 | 76 | 144 | 145 | 73
Participants
  Number of subjects with any Solicited AE | 9 | 8 | 5 | 1 | 2 | 2
  Any Solicited Local AE: number analyzed (Participants) | 144 | 145 | 73 | 144 | 145 | 73
  Any Solicited Local AE | 1 | 2 | 3 | 0 | 0 | 0
  Tenderness | 1 | 1 | 3 | 0 | 0 | 0
  Swelling/Induration | 0 | 1 | 0 | 0 | 0 | 0
  Any Solicited Systemic AE | 8 | 6 | 3 | 1 | 2 | 2
  Irritability | 1 | 0 | 1 | 0 | 0 | 0
  Drowsiness | 1 | 0 | 0 | 0 | 0 | 0
  Decrease eating | 4 | 2 | 2 | 0 | 0 | 0
  Vomiting | 3 | 4 | 0 | 1 | 1 | 1
  Fever | 4 | 2 | 3 | 0 | 1 | 2

7. Secondary Outcome: Adverse Events
Description: Unsolicited AEs reported during 28 days after each vaccination (Days 0-27 and Days 84-111);
Time Frame: 112 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Non-adjuvanted NmCV-5 (Days 0-27); Non-adjuvanted NmCV-5 (Days 84-111): Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Non-adjuvanted study formulation NmCV-5: Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysaccharide antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
- Adjuvanted NmCV-5 (Days 0-27); Adjuvanted NmCV-5 (Days 84-111): Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Adjuvanted study formulation NmCV-5: Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysaccharide antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
- Menactra (Days 0-27); Menactra (Days 84-111): Subjects in this arm will receive licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Dose to be administered is 0.5 mL intramuscularly in a two dose series separated by atleast 84 days.
  Menactra: Menactra is available as ready to used solution containing polysaccharide antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
Arm/Group | Non-adjuvanted NmCV-5 (Days 0-27) | Adjuvanted NmCV-5 (Days 0-27) | Menactra (Days 0-27) | Non-adjuvanted NmCV-5 (Days 84-111) | Adjuvanted NmCV-5 (Days 84-111) | Menactra (Days 84-111)
Number analyzed (Participants) | 149 | 150 | 76 | 144 | 145 | 73
Participants
  At least one Unsolicited AE | 37 | 39 | 23 | 23 | 17 | 16
  At least one related Unsolicited AE: number analyzed (Participants) | 144 | 145 | 73 | 144 | 145 | 73
  At least one related Unsolicited AE | 2 | 0 | 0 | 0 | 0 | 0
  At least one serious unsolicited AE | 0 | 0 | 0 | 0 | 0 | 0
  At least one serious related unsolicited AE | 0 | 0 | 0 | 0 | 0 | 0
  Unsolicited AEs leading to withdrawal from Study | 0 | 0 | 0 | 0 | 0 | 0
  Unsolicited AEs leading to withdrawal from study vaccination but remaining in the study | 0 | 0 | 0 | 0 | 0 | 0
  unsolicited AEs leading to hospitalization | 0 | 0 | 0 | 0 | 0 | 0
  Unsolicited AEs leading to Death | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Other Adverse Events
Description: AEs leading to premature withdrawal during the entire study period;
Time Frame: 168 Days
Measure: Number; unit: Number of events
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 149 | 150 | 76
Number of events | 1 | 1 | 1

9. Secondary Outcome: Serious Adverse Events
Description: SAEs reported during the entire study period
Time Frame: 168 Days
Measure: Number; unit: Number of events
Arm/Group | Non-adjuvanted Study Formulation NmCV-5 | Adjuvanted Study Formulation NmCV-5 | Menactra
Number analyzed (Participants) | 149 | 150 | 76
Number of events | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: Safety assessment includes occurrence of solicited local and systemic adverse reactions within 7 days of each vaccine dose; unsolicited adverse events within 28 days after each vaccine dose, AEs leading to withdrawal and SAE throughout the entire study period (168 days).
Groups:
- Non-adjuvanted NmCV-5 Dose 1: Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  First dose to be administered is 0.5 mL intramuscularly.
  Non-adjuvanted study formulation NmCV-5: Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
- Adjuvanted NmCV-5 Dose 1: Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  First dose to be administered is 0.5 mL intramuscularly.
  Adjuvanted study formulation NmCV-5: Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
- Menactra Dose 1: Subjects in this arm will receive licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  First dose to be administered is 0.5 mL intramuscularly. Menactra: Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
- Non-adjuvanted NmCV-5 Dose 2: Subjects in this arm will receive non-adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Second dose to be administered is 0.5 mL intramuscularly at least 84 days after Non-adjuvanted study formulation NmCV-5 Dose 1.
  Non-adjuvanted study formulation NmCV-5: Non-adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine.
- Adjuvanted NmCV-5 Dose 2: Subjects in this arm will receive adjuvanted formulation of polyvalent conjugated vaccine against meningococcal serogroups A,C,Y,W & X.
  Second dose to be administered is 0.5 mL intramuscularly at least 84 days after adjuvanted study formulation NmCV-5 dose 1.
  Adjuvanted study formulation NmCV-5: Adjuvanted formulation of polyvalent conjugate meningococcal vaccine against serogroups A,C,Y,W&X (NmCV-5) is available as lyophilised powder of polysacchride antigens A&X conjugated to tetanus toxoid and C,Y&W conjugated to CRM protein. The diluent contains Alum as adjuvant with Normal Saline. Each antigen content is 5 micrograms per 0.5 mL dose of vaccine
- Menactra Dose 2: Subjects in this arm will receive licensed quadrivalent conjugated vaccine against meningococcal serogroups A,C,Y, & W viz. Menactra.
  Second dose to be administered is 0.5 mL intramuscularly at least 84 days after Menactra dose 1.
  Menactra: Menactra is available as ready to used solution containing polysacchride antigens A,C,Y&WX conjugated to diphtheria toxoid. Each antigen content is 4 micrograms per 0.5 mL dose of vaccine.
Arm/Group | Non-adjuvanted NmCV-5 Dose 1 | Adjuvanted NmCV-5 Dose 1 | Menactra Dose 1 | Non-adjuvanted NmCV-5 Dose 2 | Adjuvanted NmCV-5 Dose 2 | Menactra Dose 2
All-Cause Mortality (participants affected / at risk) | 1/149 | 1/150 | 0/76 | 0/144 | 0/145 | 1/73
Serious Adverse Events (participants affected / at risk) | 1/149 | 1/150 | 0/76 | 0/144 | 0/145 | 1/73
Other Adverse Events (participants affected / at risk) | 41/149 | 44/150 | 25/76 | 24/144 | 17/145 | 16/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-adjuvanted NmCV-5 Dose 1 (N=149) | Adjuvanted NmCV-5 Dose 1 (N=150) | Menactra Dose 1 (N=76) | Non-adjuvanted NmCV-5 Dose 2 (N=144) | Adjuvanted NmCV-5 Dose 2 (N=145) | Menactra Dose 2 (N=73)
Escheria Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-adjuvanted NmCV-5 Dose 1 (N=149) | Adjuvanted NmCV-5 Dose 1 (N=150) | Menactra Dose 1 (N=76) | Non-adjuvanted NmCV-5 Dose 2 (N=144) | Adjuvanted NmCV-5 Dose 2 (N=145) | Menactra Dose 2 (N=73)
Injection Site Tenderness (General disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection Site Swelling/Induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowsiness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decrease Eating (General disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (General disorders) | 3 (3) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fever (General disorders) | 4 (4) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 9 (9) | 5 (5) | 7 (7) | 7 (7) | 4 (4) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Impetigo (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10) | 5 (5) | 7 (7) | 1 (1) | 5 (5)
Pharyngitis (Infections and infestations) | 10 (10) | 11 (12) | 1 (1) | 4 (4) | 5 (5) | 1 (1)
Rhinitis (Infections and infestations) | 8 (8) | 11 (12) | 7 (8) | 1 (1) | 2 (2) | 3 (3)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03295318/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/18/NCT03295318/SAP_001.pdf